CLINICAL TRIAL: NCT00439218
Title: Phase I/IIa Clinical Trial of Sodium Phenylbutyrate in Pediatric Subjects With Type I Spinal Muscular Atrophy
Brief Title: Clinical Trial of Sodium Phenylbutyrate in Children With Spinal Muscular Atrophy Type I
Acronym: NPTUNE 02
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Extremely slow enrollment
Sponsor: Westat (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: René Gonin, PhD (Math. Stats.), Senior Biostatistician and NPTUNE Principal Investigator, Westat
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01NS42361_NPTUNE02; HHSN265200423611C (Other Grant/Funding Number: NIH Contract); N01NS42361 (NIH)
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2010-07-20 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2009-05

CONDITIONS: Spinal Muscular Atrophy Type I
Keywords: spinal muscular atrophy type I; SMA type I; spinal muscular atrophy; SMA; sodium phenylbutyrate; motor neuron disease; neuromuscular; survival motor neuron; SMN; dose escalation
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal; Motor Neuron Disease | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subject Enrollments (Experimental): Cohorts of 3 subjects were to be enrolled sequentially in escalating dosage levels. The first three subjects enrolled at 500 mg/kg/day for the duration of the study drug period. The dosage of the next cohort was determined by the Modified Continual Re-assessment Method (MCRM) approach and approval of the Study Monitoring Committee (SMC). The MCRM calculation could indicate that additional subjects should be enrolled at the same dosage or a higher dosage.
  Interventions: Drug: sodium phenylbutyrate

INTERVENTIONS:
Drug: sodium phenylbutyrate — 500 mg/kg/day, depending upon tolerability subsequent dosages may increase to 675, 900, or 1200 mg/kg/day to identify maximum tolerated dose (MTD) and then an additional 6 participants will enroll at the MTD.

SUMMARY:
The purpose of this study is to identify the maximum tolerated dosage of sodium phenylbutyrate in children with spinal muscular atrophy type I; and to determine if the drug has an effect on SMN mRNA and protein levels.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a genetic, neuromuscular disorder caused by progressive degeneration of motor neurons in the spinal cord, which results from the loss of survival motor neuron (SMN) protein. The disorder is characterized by weakness and wasting of the voluntary muscles and is a leading cause of hereditary infant death. Sodium phenylbutyrate-a drug used to treat urea cycle disorders-may increase the amount of SMN protein in the body and consequently may decrease the severity of SMA. However, this has not yet been proven.

In this multicenter trial, physicians will evaluate multiple dosage levels of sodium phenylbutyrate to determine the maximum tolerated dose (MTD), or the highest dose that can be safely given to children with SMA type I. The initial dosage tested will be 500 mg/kg/day. Depending upon tolerability, subsequent groups may receive dosages of 675, 900, or 1200 mg/kg/day. Blood levels of SMN mRNA and protein will also be measured to determine whether sodium phenylbutyrate can increase the amount of these two biomarkers in the blood. Up to 24 children will be enrolled in the study, and will be on sodium phenylbutyrate for 12 weeks. The MTD will be determined based on safety data from Day 0 through the Day 29 visit. Participants will continue to be monitored for safety and SMN mRNA and protein levels through the 12 week study drug administration period.

Potential participants will be screened by having their complete medical and treatment histories recorded, as well as undergoing a physical examination, laboratory tests, and an electrocardiogram (EKG). Parents of eligible participants will receive a supply of sodium phenylbutyrate and instructions on how to administer the drug. Participants will return to the clinic on days 8, 22, 29, and at weeks 8 and 12 of the study to update their medical and treatment histories, have a physical exam, and have blood and urine collected for laboratory testing. A follow-up clinic visit will occur approximately 14 days after the last dose of sodium phenylbutyrate is given. During this visit participants will update their complete medical and treatment histories and have a physical examination. Duration of the study is about 14 weeks.

Information from this study, which is part of the NINDS Pilot Therapeutics Network (NPTUNE), may be used for future studies to determine if sodium phenylbutyrate is effective for treating SMA, and if the drug has an effect on SMA symptoms.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria within 14 days prior to receiving the first dose of study drug.

* Weakness and hypotonia consistent with a clinical diagnosis of spinal muscular atrophy (SMA) type I
* Laboratory documentation of homozygous absence of SMN1 exon 7
* Older than two months of age, but younger than 48 months of age, at the time of enrollment. If the subject is older than 24 months of age at the time of enrollment, the subject must require ventilatory support for at least 6 hours/day.
* Written informed consent of parents/guardian
* Weight greater than or equal to 7 kilograms
* Laboratory results drawn within 14 days prior to start of study drug demonstrating: Hemoglobin within normal range at the clinical site; White Blood Cell Count ≥ 3000/mm³; Platelet Count ≥ 75,000/mm³; Lipase and Amylase ≤ 1.5 x upper limit of normal (ULN) in the absence of associated clinical symptoms; AST and ALT ≤2.5x ULN; Bilirubin ≤ 1.5x ULN in the absence of associated clinical symptoms; Sodium ≥ 130 and ≤ 150 mmol/L; Potassium ≥3.0 and ≤ 5.5 mmol/L; Chloride ≤ 110 mmol/L; Calcium ≥ 8.0 mg/dL; Bicarbonate ≥ 16 mmol/L; Glucose ≥ 55 and ≤ 160 mg/dL; BUN ≤ 39 mg/dL; Creatinine ≤ 1.5 x ULN
* Subjects who are on ventilators may enroll in the protocol providing they have been on stable ventilator settings for at least the prior two weeks.
* Subject is expected to survive for at least 6 months following study entry

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participating in the study:

* Evidence of renal dysfunction, blood dyscrasia, hepatic insufficiency, symptomatic pancreatitis, cardiac arrhythmia, congenital heart defect, known history of metabolic acidosis, hypertension, significant central nervous system impairment, or neurodegenerative or neuromuscular disease other than SMA.
* Any adverse event ≥ Grade 3 at the time of screening based on the protocol toxicity grading table
* Any acute co-morbid condition interfering with the well-being of the subject within 7 days of enrollment including bacterial infection, viral infectious process, food poisoning, temperature > 99.0ºF, need for acute treatment or observation due to any other reason, as judged by the investigator.
* ≥ Grade 2 vomiting;
* ≥ Grade 2 liver dysfunction/failure (clinical);
* Any abnormality noted on EKG except for asymptomatic sinus arrhythmia
* History of allergy/sensitivity to sodium phenylbutyrate
* Use of sodium phenylbutyrate within 30 days of study entry
* Serious illness requiring systemic treatment and/or hospitalization within 14 days prior to study entry (Subjects are not eligible following serious illness until therapy is complete and the subject is stable, or until the subject is on therapy and stable for at least 14 days.)
* Poor respiratory status which is expected to require the initiation of BiPAP during the initial 29 days of drug administration.
* Use of medications intended for the treatment of SMA including riluzole, valproic acid, hydroxyurea, oral use of albuterol, sodium phenylbutyrate, butyrate derivatives, creatine, carnitine, growth hormone, anabolic steroids, probenecid, oral or parenteral use of corticosteroids at entry, haloperidol, agents anticipated to increase or decrease muscle strength or agents with known or presumed histone deacetylase (HDAC) inhibition within 30 days prior to study entry.

Notes: Subjects who use a nebulizer or require an inhaler to receive albuterol will be allowed in the study; however oral use of albuterol is prohibited. Topical use of steroids will be allowed. Oral use of steroids is not allowed at entry, but these may be used as clinically indicated while on study. Event grading will be based on the toxicity-grading table in the protocol.

Ages: 2 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: René Gonin, PhD, Principal Investigator — Mathematical Statistician, Westat; Peter R Gilbert, ScM, Study Director — The National Institute of Neurological Disorders and Stroke
Locations (5):
- United States (5):
  - Stanford University Medical Center, 300 Pasteur Drive, Room A343, Stanford, California
  - Children's Hospital, Boston, 300 Longwood Avenue, Fegan 11, Boston, Massachusetts
  - Columbia University, 180 Fort Washington Avenue, 5th Floor, New York, New York
  - The Children's Hospital of Philadelphia, Clinical Trials Office, A-230, 34th St. and Civic Center Boulevard, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Division of Pediatric Neurology, Children's Medical Center of Dallas, Ambulatory Care Pavilion, 2350 Stemmons Freeway, Suite #5074, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was open for recruitment between January 31, 2007 and April 2, 2009 at neurology clinics affiliated with university hospitals.
Pre-assignment Details: Pre-specified dosage levels of sodium phenylbutyrate(NaPB) were calculated using the modified Fibonacci rule yielding the dosage levels of 500, 675, 900 and 1200 mg /kg/day. The selection of 500 mg/kg/day as the initial dosage was based on the recommended dosage of 450 -600 mg/kg/day for the approved indication for urea cycle disorders in children.
Groups:
- Subject Enrollments: Cohorts of 3 subjects were to be enrolled sequentially in escalating dosage levels. The first three subjects enrolled at 500 mg/kg/day for the duration of the study drug period. The next cohort's dosage was determined by the Modified Continual Re-assessment Method (MCRM) approach and approval of the Study Monitoring Committee (SMC). The MCRM calculation could indicate that additional subjects should be enrolled at the same dosage or a higher dosage. Due to the replacement of a subject (1 not completed), more than 3 subjects were enrolled in cohort 1. One new subject was enrolled in Cohort 2.
Period: Cohort 1 (500 mg/kg/Day)
Arm/Group | Subject Enrollments
Started | 4
Completed | 3 (3 subjects completed the study in Cohort 1. Cohort 2 was then opened for new enrollments.)
Not Completed | 1
Not completed — Less than 80% study drug compliance | 1
Period: Cohort 2 (500 mg/kg/Day)
Arm/Group | Subject Enrollments
Started | 1 (One new subject was enrolled into the study after Cohort 1 completed the study.)
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Subject Enrollments (Cohort 1, Cohort 2): Cohorts of 3 subjects were to be enrolled sequentially in escalating dosage levels. The first three subjects enrolled at 500 mg/kg/day for the duration of the study drug period. The next cohort's dosage was determined by the Modified Continual Re-assessment Method (MCRM) approach and approval of the Study Monitoring Committee (SMC). The MCRM calculation could indicate that additional subjects should be enrolled at the same dosage or a higher dosage. Due to the replacement of a subject (1 not completed), more than 3 subjects were enrolled in cohort 1. One new subject was enrolled in Cohort 2.
Arm/Group | Subject Enrollments (Cohort 1, Cohort 2)
Number analyzed (Participants) | 5
Age, Customized [Number; unit: months]
  7-12 months | 2
  13-18 months | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLT)
Description: Number of DLTs to determine the maximum tolerated dosage. A DLT is defined as any Grade(GR)3 or higher adverse event, GR 1 or higher cardiac arrhythmia; GR 2 or higher vomiting; GR 2 or higher liver dysfunction/failure (clinical); GR 2 elevation of amylase or lipase accompanied by clinical symptoms of pancreatitis. The following GR 2 events are classified as DLTs if evaluated to be clinically significant by the principal investigator or medical safety monitor: decrease of hemoglobin, WBCs, platelets; elevation of AST, ALT, bilirubin; abnormlity of Na, K, Cl, CA, HCO3, glucose, BUN, creatinine.
Time Frame: 29 days
Population: The study was closed prematurely due to slow accrual. The MTD could not be determined due to the small number of subjects enrolled.
Measure: Number; unit: DLT(s)
Arm/Group | Subject Enrollments
Number analyzed (Participants) | 0

2. Primary Outcome: Survival Motor Neuron (SMN) Messenger Ribonucleic Acid (mRNA)
Description: The change of level in blood SMN mRNA from baseline to assess time course and dose response.
Time Frame: Baseline - 12 weeks
Population: The study was closed prematurely due to slow accrual. These data are exploratory and have not yet been analyzed. Their interpretability will be limited because of the small number of specimens collected.
Measure: Mean (Standard Error); unit: Cycle Threshold (Ct)
Arm/Group | Subject Enrollments
Number analyzed (Participants) | 0

3. Secondary Outcome: Drug Safety
Description: Adverse event (AE) monitoring
Time Frame: 14 weeks
Population: The study was closed prematurely due to slow accrual. These data have not yet been analyzed. Their interpretability will be limited because of the small number of subjects enrolled. There were no safety concerns reported by the SMC.
Measure: Number; unit: Adverse Events
Arm/Group | Subject Enrollments
Number analyzed (Participants) | 0

4. Primary Outcome: Survival Motor Neuron (SMN) Protein
Description: The change of level in blood SMN protein from baseline to assess time course and dose response.
Time Frame: Baseline - 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SMN/beta tubulin
Arm/Group | Subject Enrollments
Number analyzed (Participants) | 0

5. Secondary Outcome: Pharmacokinetic Parameters (Maximum Plasma Concentration)
Description: Maximum Plasma Concentration (Cmax)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Subject Enrollments
Number analyzed (Participants) | 0

6. Secondary Outcome: Pharmacokinetic Parameters (Time to Maximum Plasma Concentration)
Description: Time to maximum plasma concentration (Tmax)
Time Frame: 12 weeks
Population: The study was closed prematurely due to slow accrual. These data have not yet been analyzed. Their interpretability will be limited because of the small number of specimens collected.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Subject Enrollments
Number analyzed (Participants) | 0

7. Secondary Outcome: Pharmacokinetic Parameters (Area Under the Plasma Concentration Versus Time Curve (AUC))
Description: Area under the plasma concentration versus time curve (AUC)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: µmol/L * hours
Arm/Group | Subject Enrollments
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Study Drug Compliance
Description: Subjects receiveing 80% or more of the prescribed doses within each study visit interval were considered compliant.
Time Frame: 12 weeks
Population: A total of 5 participants were enrolled in the study. Four enrolled in Cohort 1.
Measure: Number; unit: Participants
Arm/Group | Subject Enrollments
Number analyzed (Participants) | 5
Participants
  Cohort 1 (500 mg/kg/day) | 3
  Cohort 2 (500 mg/kg/day) | 1

ADVERSE EVENTS:
Time Frame: Data were collected over a 2 year period.
Description: Data were collected at scheduled clinic and telephone study visits via medical history, physical examinations, laboratory tests, EKG, and other tests as necessary. In addition, adverse events were reported to site investigators by subjects' parents in between visits, as needed.
Arm/Group | Subject Enrollments
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject Enrollments (N=5)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject Enrollments (N=5)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Eye movement disorder (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Saliva altered (Gastrointestinal disorders) | 1 (1)
Teething (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Pyrexia (General disorders) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Otitis Media (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
AST increased (Investigations) | 3 (3)
Blood bicarbonate increased (Investigations) | 1 (1)
Blood chloride increased (Investigations) | 2 (2)
Blood urine present (Investigations) | 1 (2)
Glucose urine present (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertonia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was closed early due to slow accrual. The sample size is therefore extremely limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must submit an application to the NPTUNE Publications Committee for the use of data. A Writing Committee, appointed by the Publications Committee, is responsible for initiating, coordinating, and approving publications and presentations.